CLINICAL TRIAL: NCT00918190
Title: Late Onset Postoperative Nausea and Vomiting Following Strabismus Surgery in Pediatric.What Combination is Better
Brief Title: Late Onset Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khaled Eye Specialist Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RP 0917
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative nausea and vomiting; Pediatric; Strabismus; Late onset postoperative nausea and vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Strabismus; Vomiting | interventions — Sodium Chloride; Ondansetron; Dexamethasone; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ondansetron-Dexa group (Active Comparator): Use 2 different antiemetics
  Interventions: Drug: Ondansetron, Dexamethasone
- Midazolam, Dexa group (Active Comparator): use of midazolam and dexamethasone
  Interventions: Drug: Midazolam, dexamethasone
- Placebo (Placebo Comparator): Saline will be given
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Saline
  Other Names: saline
  Arms: Placebo
Drug: Ondansetron, Dexamethasone — Use of ondansetron and dexamethasone as combined antiemetics
  Other Names: Zofran
  Arms: Ondansetron-Dexa group
Drug: Midazolam, dexamethasone — use of midazolam and dexamethasone as combined antiemetic
  Other Names: Midazolam
  Arms: Midazolam, Dexa group

SUMMARY:
The purpose of this trial is to study the effects of different combinations of antiemetics on the incidence of late onset postoperative nausea and vomiting.

DETAILED DESCRIPTION:
The authors will study the effect of many antiemetics on the occurrence of nausea and vomiting following strabismus surgery in pediatrics.

ELIGIBILITY:
Inclusion Criteria:

* children undergoing elective strabismus surgery under general anesthesia

Exclusion Criteria:

* children experienced retching or vomiting
* children who have taken anti-emetic medications, antihistaminics, steroids, or psychoactive drugs within 24 hours before surgery

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of antiemetics combination | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Riad, MD, AB, SB, Principal Investigator — King Khaled Eye Specialist Hospital
Locations (1):
- king Khaled Eye Specialist hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Riad W, Altaf R, Abdulla A, Oudan H. Effect of midazolam, dexamethasone and their combination on the prevention of nausea and vomiting following strabismus repair in children. Eur J Anaesthesiol. 2007 Aug;24(8):697-701. doi: 10.1017/S0265021507000166. Epub 2007 Apr 17. PMID 17437654